CLINICAL TRIAL: NCT00244114
Title: In Vitro Evaluation Of Allergic Reactions In Hemophilia B Subjects Who Have Exhibited A Systemic Allergic Response After Exposure To BeneFIX (Nonacog Alfa; Recombinant Factor IX)
Brief Title: Study Evaluating Allergic Reactions To Benefix In Hemophilia B Patients
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3090A1-900; B1821003; 3090A-101795
Record Dates: First submitted 2005-10-19; First posted 2005-10-25 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Allergic Reaction
MeSH Terms: conditions — Hemophilia B; Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: blood draw
- B
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Drug: blood draw — Single blood sample collected to perform histamine release assay.
  Groups: A
Procedure: Blood draw — Single blood sample collected to perform histamine release assay.
  Groups: B

SUMMARY:
Based on the finding that anaphylactic reactions to Benefix ("FIX") are associated with a specific IgE, a Basophil histamine release assay was selected to evaluate and demonstrate subject sensitization to FIX.

ELIGIBILITY:
Inclusion Criteria:

Study Group:

* Written informed consent or assent, as applicable.
* Subjects with moderate to severe Hemophilia B (FIX:C <5%), who have reported class II or class III allergic manifestations within 24 hours of a BeneFIX infusion.

Control Group:

* Written informed consent or assent, as applicable.
* Subjects with moderate to severe Hemophilia B (FIX:C <5%)

Exclusion Criteria:

Study group:

* Subjects who had no reaction when rechallenged with BeneFIX, in the absence of prophylactic immunomodulating therapy.
* Subjects whose most recent allergic manifestations with BeneFIX occurred >36 months prior to providing written informed consent for this study.
* Subjects who have taken antihistamine, steroidal, or other immunosuppressive therapy within 72 hours of the scheduled visit for this study.
* Subjects with immune disorders.
* Subjects unable to comply with a minimum 5-day FIX washout requirement.

Control group:

* Subjects with documented evidence of prior allergic reaction to any FIX product.
* Subjects with documented evidence of prior or current FIX inhibitor (BU >0.6).
* Subjects have taken antihistamine, steroidal, or other immunosuppressive therapy within 72 hours of the scheduled study blood draw.
* Subjects with immune disorder.
* Subjects unable to comply with a minimum 5-day FIX washout requirement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Descriptive presentation of the results of the Basophil histamine release assay for both study and control groups | within 36 months after allergic reaction

SECONDARY OUTCOMES:
Collect and evaluate adverse events that occur from the time the subject signs the informed consent form to 15 days following the study visit will be collected | 15 days
Any serious adverse events and/or adverse events of special interest occurring outside of the predefined study reporting period noted to be possibly, probably or definitely related to treatment with BeneFIX will be reported. | 15 days following study blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090A1-900&StudyName=Study%20Evaluating%20Allergic%20Reactions%20To%20Benefix%20In%20Hemophilia%20B%20Patients